CLINICAL TRIAL: NCT05249075
Title: Micro-Tech FNB Needle to Obtain Tissue Specimens of Pancreas Malignancy for Personalized Based Chemotherapy
Acronym: MT-FNB
Status: Active, not recruiting | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 112922
Record Dates: First submitted 2022-02-10; First posted 2022-02-21 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Systemic chemotherapy can improve disease-related symptoms and/or prolong survival in patients with pancreatic cancer. Before the start of chemotherapy, the diagnosis pancreatic carcinoma must be confirmed by tumor tissue samples, which are often obtained during endoscopic ultrasound (EUS) by fine needle aspiration (FNA) or fine needle biopsy (FNB). Obtaining core biopsies by FNB has several potential benefits, such as making a more reliable diagnosis, performing immunohistochemistry for diagnostic reasons and in the future obtaining enough malignant cells to deliver personalized based chemotherapy regimen based on mutations detected by next generation sequencing. Obtaining high quality and sufficient tumor material is essential for genomic profiling with a preference of FNB over FNA. Up to now, no specific FNB needle has been found to be superior in diagnostic accuracy and in obtaining tissue for genomic profiling. In this study, we aim to evaluate the diagnostic accuracy of a new FNB needle (Micro-Tech Europe GmbH, Düsseldorf, Germany) and we study the adequacy of the obtained tissue samples for performing genetic sequencing.

DETAILED DESCRIPTION:
This study is an international multicenter prospective cohort study. The study will be performed in collaboration with the disciplines of Gastroenterology and Pathology of the participating hospitals.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Clinical suspicion of pancreatic adenocarcinoma
* Indication for obtaining EUS-guided histology of a suspected pancreatic lesion
* Written informed consent

Exclusion Criteria:

* Contra-indications to undergoing an EUS (e.g., oropharyngeal abnormalities)
* Altered anatomy (e.g., after previous Whipple-operation, Roux-and-Y gastrojejunostomy)
* Contra-indications to the administration of benzodiazepines, propophol or opioids
* Pregnancy
* Insufficient knowledge of the Dutch language to be able to understand the patient information

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Each patient with clinical suspicion of pancreatic cancer, based on imaging, will be discussed in the multidisciplinary team consultation. When an EUS-FNB is indicated, patients are included if they meet all the inclusion and none of the exclusion criteria.
  The population will consist of elderly patients, as pancreatic cancer is rarely diagnosed before the age of 55.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2025-08-14 (Actual); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of the Micro-Tech FNB needle in obtaining pancreatic malignancy | 2 years
  Pathologist scores the obtained specimen according the Bethesda system. Diagnostic accuracy will be quantified by the sensitivity and specificity and expressed as frequency of pancreatic malignancy as confirmed by histological evaluation.

SECONDARY OUTCOMES:
Ability to perform genetic sequencing on the sample | 2 years
  Pathologist will analyze the obtained specimen and determines the size and tumor cellularity. The specimen is deemed sufficient for performing genetic sequencing when tumor cellularity is >20% and the surface is >5mm2. At this stage, no genetic sequencing will be performed
Puncture success rate | 2 years
  Puncture is successful if the pathologist is able to make a diagnosis on the obtained specimen. By putting each biopsy in a different formalin jar, we can count how many biopsies are needed to be taken to obtain a representative biopsy for diagnosis.
User experience | 2 years
  User experience of performing FNB with this needle scored with a questionnaire filled in by each participating gastroenterologist after performing all procedures.

CONTACTS AND LOCATIONS:
Overall Officials: Erwin van Geenen, MD, PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboudumc, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
The dataset used during this study is available from the corresponding author upon reasonable request.